CLINICAL TRIAL: NCT03842657
Title: Regional Anticoagulation of Dialysis Extra-corporeal Circuits With a Calcium-free Citrate-containing Dialysate : Efficiency and Tolerance
Brief Title: Regional Anticoagulation of Dialysis Circuits With a Calcium-free Citrate-containing Dialysate
Acronym: C2D
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RC31/17/0451
Record Dates: First submitted 2019-01-29; First posted 2019-02-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2022-03

CONDITIONS: Hemodialysis Complication; Bleeding
Keywords: citrate, dialysate; hemodialysis; coagulation
MeSH Terms: conditions — Hemorrhage; Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- calcium-free citrate-containing dialysate (Other): Dialysis session will be performed with a non-heparin grafted membrane, a dialysate without calcium (0 mmol/L) and citrate 0.8 mmol/L, a reinjection of a calcium solution (300 mM) according to the ionic dialysance, and no heparin addition
  Interventions: Combination Product: anticoagulation of the dialysis circuit
- heparin-grafted membrane (Other): dialysis session will be performed with a heparin-grafted membrane, a dialysate with calcium (1.65 mmol/L) and citrate 0.8 mmol/L, and no heparin addition
  Interventions: Combination Product: anticoagulation of the dialysis circuit

INTERVENTIONS:
Combination Product: anticoagulation of the dialysis circuit — Each patient included in this study will receive two heparin-free dialysis sessions with heparin-grafted membrane (control group) or RCA with calcium-free citrate-containing dialysate and calcium reinjection according to the ionic dialysance (experimental group), alternatively

SUMMARY:
Critically ill patients have a high risk of bleeding but also require prolonged intermittent dialysis. Thus, a heparin-free easy-to-use alternative type of anticoagulation within the dialysis circuit is required. In a non-comparative study, heparin-free regional citrate anticoagulation of the dialysis circuit using a calcium-free citrate-containing dialysate, with calcium reinjected according to ionic dialysance, was considered as safe and efficient. The aim of this study is to confirm the superiority of this approach compared to a anticoagulation based on heparin-grafted membrane.

DETAILED DESCRIPTION:
Critically ill patients have a high risk of bleeding but also require prolonged intermittent dialysis. Several modalities are used for heparin-free dialysis sessions. Iterative saline infusion and heparin-grafted membranes are easy to use and remain the standards-of-care for high-risk bleeding situations but efficiency is low: success rates from hemodialysis sessions range from 50% to 65% and 50% to 75%, respectively. Furthermore, sessions that last for greater than 240 minutes are rarely achievable and can be problematic when ensuring an adequate dose of dialysis and a negative water balance in patients who cannot tolerate a high ultrafiltration rate. Thus, the development of alternative regional anticoagulation methods is needed urgently to improve intermittent hemodialysis (IHD) in critically ill patients and to avoid systemic anticoagulation in patients with a high risk of bleeding.

An easy way to provide citrate inside the filter, to lower iCa below 0.45 mmol/L could be to use diffusive influx from the dialysate. It has been demonstrated recently that the use of citric acid as the acidic component of dialysate can enable a dose reduction of heparin and increase the efficiency of hemodialysis. However, the amount of citrate (0.8 mmol/L) and calcium (1.25-1.75 mmol/L) contained in this dialysate do not allow the target of iCa to be reached in the ECC. In contrast, a citrate dialysate that contains no calcium would provide enough calcium-free transfer to lower iCa below 0.45 mmol/L; however, a problem would be the large amount of calcium loss during the session.

Pivotal studies show that, during dialysis sessions performed with calcium-free dialysate, the rate of calcium reinjection required to compensate for calcium loss in the dialysate can be easily deducted from the ionic dialysance (ID), which is an online measurement of instantaneous small solute clearance, available from most dialysis monitors. ID has been also used as a surrogate marker for dialysis dose in ICU patients receiving IHD. Thus, the use of calcium-free citrate-containing dialysate with calcium reinjection according to ID could provide enough citrate to prevent coagulation within the filter, and calcium restitution can then be monitored by online ID without the need for systemic measurement of iCa. It may also improve the hemodynamic tolerance of IHD by avoiding acetate in the dialysate.

The objective of the present study was to show the efficiency of this approach using RCA for dialysis sessions (<4 hrs) of IHD in patients with moderate to high risk of bleeding, based on the success rate of hemodialysis without clotting. Each patient included in this study will receive two heparin-free dialysis sessions with heparin-grafted membrane (control group) or RCA with calcium-free citrate-containing dialysate and calcium reinjection according to the ionic dialysance (experimental group), alternatively. The order of anticoagulation will be randomized.

ELIGIBILITY:
Inclusion Criteria: will be included in the study, patients

* hat require two sessions of dialysis that last for greater than 240 minutes in the 7 days following the inclusion.
* With a moderate to high risk of bleeding (platelets count below 150.000/mm3; platelet disorders; bleeding in the last 10 days, surgery or biopsy in the last 10 days or planned in the next 7 days; admission to the ICU)
* Older than 18 years of age
* That gave written informed consent

Exclusion Criteria: will be excluded from the study, patients with

* Heparin allergy
* On-going treatment by vitamin-K antagonists (INR > 1.2) or unfractionated heparin (anti-Xa activity > 0.10)..
* Known allergy to the Evodial (Baxter, France) or Cordiax FX100 (Fresenius, France) membranes
* On-going treatment by angiotensin converting enzyme inhibitors
* Pregnancy or risk of pregnancy
* Patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2021-09-13 (Actual)

PRIMARY OUTCOMES:
Premature termination of the first dialysis session (<4 hours) related to a coagulation of the dialysis circuit | Visite T1 (3 days maximum after inclusion visit)
  Premature termination of the dialysis session (<4 hours) in connection with coagulation or pre-coagulation state of the dialysis circuit (thrombosis global index strictly greater than 1 (visual assessment) or elevation of transmembrane pressure above 350 mmHg)
Premature termination of the second dialysis session (<4 hours) related to a coagulation of the dialysis circuit | Visite T2 (7 days maximum after inclusion visit)
  Premature termination of the dialysis session (<4 hours) in connection with coagulation or pre-coagulation state of the dialysis circuit (thrombosis global index strictly greater than 1 (visual assessment) or elevation of transmembrane pressure above 350 mmHg)

SECONDARY OUTCOMES:
Hemodynamic tolerance | Visite T1 (3 days maximum after inclusion visit), Visite T2 (7 days maximum after inclusion visit)
  Number of cardiovascular events during the dialysis session
Clinical tolerance | Visite T1 (3 days maximum after inclusion visit), Visite T2 (7 days maximum after inclusion visit)
  Clinical symptoms collected every 30 min on patient
Biological tolerance | Visite T1 (3 days maximum after inclusion visit), Visite T2 (7 days maximum after inclusion visit)
  Measurement of total and ionized calcium and venous pH sampled on the arterial branch of the dialysis circuit
Systemic inflammation | Visite T1 (3 days maximum after inclusion visit), Visite T2 (7 days maximum after inclusion visit)
  To determine the serum levels of cytokines (interleukine-6, interferon-γ, MCP1, Tumor Necrosis Factor-α) by ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Stanislas FAGUER, MD, Principal Investigator — University Hospital, Toulouse
Locations (5):
- France (5):
  - Pellegrin Hospital, Bordeaux
  - Montpellier Hospital, Montpellier
  - Nimes Hospital, Nîmes
  - Tenon Hospital, Paris
  - CHU Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Faguer S, Serre JE, Brusq C, Bongard V, Casemayou A, Moranne O, Pfirmann P, Rafat C, Cointault O. A randomized crossover trial of regional anticoagulation modalities for intermittent haemodialysis. Nephrol Dial Transplant. 2025 Feb 28;40(3):537-543. doi: 10.1093/ndt/gfae155. PMID 38977911